CLINICAL TRIAL: NCT01711866
Title: An Open-Label, Multicenter, Multinational Study to Assess the Feasibility of Switching Therapy From Pramipexole or Ropinirole to the Rotigotine Transdermal System and Its Effect on Motor and Non-Motor Symptoms in Subjects With Advanced Idiopathic Parkinson's Disease Phase 4
Brief Title: A Phase 4, Open-label Study to Assess the Feasibility and Efficacy on Motor and Non-motor Symptoms of Switching From Pramipexole or Ropinirole to Rotigotine Transdermal Patch in Subjects With Advanced Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD0009
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro; Switch; Dopamine agonists
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): First application of Rotigotine patch for 24 hours on Day 1, followed by application of a new patch each day of the Treatment Period.
  * Subjects on lower doses switch from Pramipexole or Ropinirole to equivalence doses of Rotigotine on Day 1 of the 28 days Treatment Period. On Day 8 (Visit 3) the dose will be evaluated and potentially adjusted up to a maximum dose of 8 mg / 24 hours.
  * Subjects on higher doses switch from the equivalent dose to 8 mg / 24 hours Rotigotine of Pramipexole or Ropinirole to 8 mg / 24 hours Rotigotine on Day 1 and the remainder of the dose of Pramipexole or Ropinirole is to be switched on Day 8 of the 28 days Treatment Period. On Day 15 (Visit 4) the dose will be evaluated and potentially adjusted up to a maximum dose of 16 mg / 24 hours.
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine up to 16 mg / 24 hours, 4 weeks.
  Other Names: Neupro

SUMMARY:
The purpose of this study is to assess the safety and feasibility of switching subjects with advanced Parkinson's Disease (PD) from Pramipexole or Ropinirole to Rotigotine and to assess the effects of Rotigotine on motor and non-motor symptoms of Parkinson's Disease in subjects switched from previous treatment with either Pramipexole or Ropinirole.

ELIGIBILITY:
Inclusion Criteria:

* Subject has idiopathic Parkinson's Disease of more than 3 years duration, as defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, impairment of postural reflexes and is without any other known or suspected cause of Parkinsonism
* Subject has motor fluctuations
* Subject is not satisfactorily controlled following the investigator´s assessment on a total daily dose of Pramipexole or Ropinirole
* Subject has sleep disturbance or early morning motor impairment
* Subject has experienced nocturia for at least 3 nights within 7 days prior to the Baseline Visit
* Subject is taking L-dopa in combination with Benserazide or Carbidopa and has been on a stable dose of L-dopa for at least 28 days prior to the Baseline Visit

Exclusion Criteria:

* Subject has had therapy with Tolcapone or Budipine
* Subject is receiving therapy with one of the following drugs either concurrently or within 28 days prior to Baseline (Visit 2): alpha-methyl dopa, metoclopramide, reserpine, neuroleptics, monoamine oxidase A (MAO-A) inhibitors, methylphenidate, or amphetamine
* Subject has a history of symptomatic (not asymptomatic) orthostatic hypotension in the 6 months prior to Baseline (Visit 2)
* Subject has a history of significant skin hypersensitivity to adhesive or other transdermal preparations, or recent unsolved contact dermatitis
* Subject has a history of seizures or stroke within 1 year, or a history of myocardial infarction within the last 6 months prior to enrollment
* Subject is pregnant or nursing, or is of childbearing potential but (i) not surgically sterile or (ii) not using adequate birth control methods (including at least 1 barrier method) or (iii) not sexually abstinent or (iv) not at least 2 years postmenopausal
* Subject has a previous diagnosis of narcolepsy, sleep apnea syndrome, restless legs syndrome, or periodic limb movement disorder

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (21):
- United States (6):
  - 505, Anniston, Alabama
  - 506, Atlantis, Florida
  - 508, Miami Springs, Florida
  - 502, Atlanta, Georgia
  - 501, Dayton, Ohio
  - 509, Oklahoma City, Oklahoma
- 202, Sarawak, Malaysia
- Singapore (2):
  - 401, Singapore
  - 403, Singapore
- South Korea (9):
  - 101, Busan
  - 102, Busan
  - 108, Daegu
  - 109, Daegu
  - 105, Gyeonggi-do
  - 103, Seoul
  - 104, Seoul
  - 106, Seoul
  - 107, Seoul
- Taiwan (3):
  - 301, Linkou District
  - 304, Taichung
  - 305, Taipei

REFERENCES:
- [Derived] Chung SJ, Kim JM, Kim JW, Jeon BS, Singh P, Thierfelder S, Ikeda J, Bauer L; Asia Pacific Rotigotine Switching Study Group. Switch from oral pramipexole or ropinirole to rotigotine transdermal system in advanced Parkinson's disease: an open-label study. Expert Opin Pharmacother. 2015 May;16(7):961-70. doi: 10.1517/14656566.2015.1030336. Epub 2015 Apr 6. PMID 25846031
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in September 2012 in order to enroll 87 subjects in 5 countries.
  Participant Flow refers to the Safety Set (SS). SS consists of all subjects who were enrolled and had at least 1 patch applied during the Treatment Period.
Groups:
- Rotigotine: First application of Rotigotine patch for 24 hours on Day 1, followed by application of a new patch each day of the Treatment Period.
  * Subjects on lower doses switch from Pramipexole or Ropinirole to equivalence doses of Rotigotine on Day 1 of the 28 days Treatment Period. On Day 8 (Visit 3) the dose will be evaluated and potentially adjusted up to a maximum dose of 8 mg / 24 hours.
  * Subjects on higher doses switch from the equivalent dose to 8 mg / 24 hours Rotigotine of Pramipexole or Ropinirole to 8 mg / 24 hours Rotigotine on Day 1 and the remainder of the dose of Pramipexole or Ropinirole is to be switched on Day 8 of the 28 days Treatment Period. On Day 15 (Visit 4) the dose will be evaluated and potentially adjusted up to a maximum dose of 16 mg / 24 hours.
  Rotigotine: Rotigotine up to 16 mg / 24 hours, 4 weeks.
Period: Overall Study
Arm/Group | Rotigotine
Started | 87
Completed | 79
Not Completed | 8
Not completed — Noncompliant | 3
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set. The Safety Set consists of all subjects who had at least one patch application.
Arm/Group | Rotigotine
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 6
  Taiwan | 9
  Malaysia | 1
  Singapore | 2
  Korea, Republic of | 69

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression (CGI) Item 4 (Side Effects) at the End of the Treatment Period or Early Withdrawal Visit
Description: The CGI Item 4 was used to assess side effects. It ranges from 0 to 4 as follows:
  * 0 = Side effects not assessable
  * 1 = No side effects
  * 2 = Side effects do not significantly interfere with subject's functioning
  * 3 = Side effects significantly interfere with the subject's functioning
  * 4 = Side effects outweigh therapeutic efficacy.
Time Frame: Day 28 (Visit 5) of the 28 days Treatment Period or Early Withdrawal Visit
Population: All 87 subjects of the Safety Set are included in the analysis of this outcome measure. Last Observation Carried Forward (LOCF) was used as a method of imputation for missing observations.
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 87
participants
  CGI Item 4 score of 1 | 58
  CGI Item 4 score of 2 | 26
  CGI Item 4 score of 3 | 3
  CGI Item 4 score of 4 | 0
  CGI Item 4 score of 3 or 4 | 3

2. Secondary Outcome: Patients Global Impressions of Change (PGIC) at the End of the Treatment Period or Early Withdrawal Visit
Description: The PGIC is a 7-point categorical rating scale in which the subject rates the changes in functioning over time as follows:
  * 1 = Very much improved
  * 2 = Much improved
  * 3 = Minimally improved
  * 4 = No change
  * 5 = Minimally worse
  * 6 = Much worse
  * 7 = Very much worse.
Time Frame: Day 28 (Visit 5) of the 28 days Treatment Period or Early Withdrawal Visit
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF) as a method of imputation for missing observations. FAS includes all subjects with at least 1 patch application during Treatment Period, and with an evaluable UPDRS Part III total score at Baseline and at least 1 valid value after Baseline to Day 35.
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 84
participants
  PGIC category 1 | 5
  PGIC category 2 | 17
  PGIC category 3 | 30
  PGIC category 4 | 18
  PGIC category 5 | 10
  PGIC category 6 | 3
  PGIC category 7 | 1
  PGIC category ≥ 5 | 14
  PGIC category ≥ 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the whole study duration from the Screening Period (Day -28 to Day -1) to the Safety Follow-up Visit (up to Day 54).
Description: Adverse Events refer to the Saftey Set. Safety Set consists of all subjects who were enrolled and had at least 1 patch applied during the Treatment Period.
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 1/87
Other Adverse Events (participants affected / at risk) | 30/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=87)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=87)
Application site pruritus (General disorders) | 9 (9)
Application site erythema (General disorders) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6)
Dyskinesia (Nervous system disorders) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days